CLINICAL TRIAL: NCT00107458
Title: A Phase I Study of Valproic Acid in Children With Recurrent/Progressive Solid Tumors Including CNS Tumors
Brief Title: Valproic Acid in Treating Young Patients With Recurrent or Refractory Solid Tumors or CNS Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ADVL0419; COG-ADVL0419 (Other: Children's Oncology Group); NCI-05-C-0235; NCI-P6631; CDR0000417845 (Other: Clinical Trials.gov)
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Brain and Central Nervous System Tumors; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: recurrent childhood brain stem glioma; recurrent childhood brain tumor; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood ependymoma; recurrent childhood medulloblastoma; recurrent childhood supratentorial primitive neuroectodermal tumor; unspecified childhood solid tumor, protocol specific; recurrent childhood visual pathway and hypothalamic glioma; childhood high-grade cerebral astrocytoma; childhood low-grade cerebral astrocytoma; childhood infratentorial ependymoma; childhood supratentorial ependymoma; childhood spinal cord neoplasm; childhood grade I meningioma; childhood grade II meningioma; childhood grade III meningioma; childhood craniopharyngioma; childhood central nervous system germ cell tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Familial ependymoma; Medulloblastoma; Optic Nerve Glioma; Spinal Cord Neoplasms | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment 1 (Experimental): VPA Target Trough Concentration 75-100 mcg/mL, week 1 VPA dose: 15 mg/kg/day, divided tid
  Interventions: Drug: valproic acid
- Treatment 10 (Experimental): VPA Target Trough Concentration 100-150 mcg/mL, week 1 VPA dose: 15 mg/kg/day, divided tid
  Interventions: Drug: valproic acid
- Treatment 20 (Experimental): VPA Target Trough Concentration 150-200 mcg/mL
  Interventions: Drug: valproic acid

INTERVENTIONS:
Drug: valproic acid

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as valproic acid, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Valproic acid may also stop the growth of solid tumors or CNS tumors by blocking blood flow to the tumor.

PURPOSE: This phase I trial is studying the side effects and best dose of valproic acid in treating patients with recurrent or refractory solid tumors or CNS tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxic effects of valproic acid (VPA) administered at doses required to maintain serum trough VPA concentrations of 100-150 mcg/mL or 150-200 mcg/mL in young patients with recurrent or refractory solid tumors or CNS tumors.

Secondary

* Determine the steady-state serum trough concentration of free and total VPA at the targeted total trough VPA concentration in these patients.
* Determine the steady state histone acetylation status of peripheral blood monocytes at the targeted trough VPA concentration in these patients.
* Determine the pharmacokinetic profile of this drug in these patients.
* Correlate histone acetylation with free or total trough VPA concentration in these patients.
* Determine, preliminarily, the antitumor activity of this drug in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

For course 1, patients receive escalating doses of oral valproic acid (VPA) twice daily until a target serum trough VPA concentration range is maintained for 28 days. Patients who achieve the target serum trough VPA concentration range receive subsequent courses of oral VPA twice daily (at the dose found to maintain the target serum trough VPA concentration range) on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

The first cohort of 6 patients receives VPA to achieve an initial target trough serum VPA concentration. If fewer than 2 of 6 patients in the first cohort experience dose-limiting toxicity (DLT), then a second cohort of 6 patients receives VPA to achieve the next higher target trough serum VPA concentration. If fewer than 2 patients from the second cohort experience DTL, then 6 additional patients are enrolled in this cohort to better define pharmacokinetics and DLT at this VPA concentration range.

After completion of study treatment, patients are followed annually.

PROJECTED ACCRUAL: A total of 12-18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed* malignant solid tumor, including CNS tumors, at original diagnosis or relapse

  * Recurrent or refractory disease NOTE: *Histologic confirmation not required for intrinsic brain stem or optic pathway tumors
* Measurable or evaluable disease, defined by 1 of the following criteria:

  * Any unidimensionally measurable lesion ≥ 10 mm by standard MRI or CT scan for either solid or CNS tumors
  * At least 1 nonmeasurable lesion that is evaluable by nuclear medicine, immunocytochemistry, tumor markers, cerebrospinal fluid cytology, or other reliable measures
* No known curative therapy exists
* No documented tumor involvement in the bone marrow

PATIENT CHARACTERISTICS:

Age

* 2 to 21

Performance status*

* Lansky 50-100% (for patients ≤ 10 years of age)
* Karnofsky 50-100% (for patients > 10 years of age)

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3 (transfusion independent)
* Hemoglobin ≥ 8.0 g/dL (transfusions allowed)

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 110 (ULN for this study is 45 U/L)
* Albumin ≥ 2 g/dL

Renal

* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR
* Creatinine based on age as follows:

  * No greater than 0.8 mg/dL (for patients ≤ 5 years of age)
  * No greater than 1.0 mg/dL (for patients 6 to 10 years of age)
  * No greater than 1.2 mg/dL (for patients 11 to 15 years of age)
  * No greater than 1.5 mg/dL (for patients over 15 years of age)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Neurologic deficits in patients with CNS tumors must be stable for ≥ 1 week before study entry
* No uncontrolled infection
* No known urea cycle disorders or other metabolic disorders
* No other condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Recovered from prior immunotherapy
* At least 7 days since prior hematopoietic growth factors that support platelet or WBC number or function
* At least 7 days since prior antineoplastic biologic agents
* At least 3 months since prior stem cell transplantation or rescue without total body irradiation

  * No evidence of active graft vs host disease
* No other concurrent anticancer biologic therapy or immunotherapy

Chemotherapy

* More than 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas) and recovered
* No other concurrent anticancer chemotherapy

Endocrine therapy

* Patients with CNS tumors must be on a stable or decreasing dose of dexamethasone for the past 7 days

Radiotherapy

* See Biologic therapy
* Recovered from prior radiotherapy
* At least 6 months since prior total body irradiation, craniospinal radiotherapy, or radiotherapy to ≥ 50% of the pelvis
* At least 6 weeks since other prior substantial bone marrow radiotherapy
* At least 2 weeks since prior local palliative small port radiotherapy
* No concurrent anticancer radiotherapy

Surgery

* Not specified

Other

* No other concurrent investigational agents
* No other concurrent anticancer agents
* No other concurrent anticonvulsants

  * Patients receiving valproic acid (VPA) before study entry must have a total trough VPA concentration < 100 mcg/mL within the past 7 days

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2005-05; Primary Completion 2007-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of oral etoposide at 50 mg/m2/day given concurrently with radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jack M. Su, MD, Study Chair — Texas Children's Cancer Center; Heidi V. Russell, MD, Study Chair — Texas Children's Cancer Center
Locations (17):
- United States (15):
  - Children's Hospital of Orange County, Orange, California
  - Stanford Comprehensive Cancer Center - Stanford, Stanford, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota Children's Hospital - Fairview, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health & Science University Cancer Institute, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor University Medical Center - Houston, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
- Canada (2):
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Sainte Justine, Montreal, Quebec

REFERENCES:
- [Result] Su JM, Li XN, Thompson P, Ou CN, Ingle AM, Russell H, Lau CC, Adamson PC, Blaney SM. Phase 1 study of valproic acid in pediatric patients with refractory solid or CNS tumors: a children's oncology group report. Clin Cancer Res. 2011 Feb 1;17(3):589-97. doi: 10.1158/1078-0432.CCR-10-0738. Epub 2010 Nov 29. PMID 21115653